CLINICAL TRIAL: NCT06321653
Title: AXILL-ART: Lymphedema Evaluation After Adjuvant Hypofractionated Radiotherapy for 1-2 Macrometastatic Sentinel Lymph Nodes Without Axillary Dissection in Breast Cancer Conservative Surgery: Observational Study
Brief Title: Lymphedema Evaluation After Adjuvant Hypofractionated Radiotherapy for 1-2 Macrometastatic Sentinel Lymph Nodes
Acronym: AXILL-ART
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 0953
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Arm Lymphedema; Breast Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypofractionated radiotherapy: Hypofractionated radiotherapy scheme with 2.67Gy/fraction for 15 fractions. WBRT with simultaneous integrated boost to the tumor bed
  Interventions: Radiation: Hypofractionated radiotherapy scheme

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy scheme — Hypofractionated radiotherapy scheme with 2.67Gy/fraction for 15 fractions. WBRT with simultaneous integrated boost to the tumor bed

SUMMARY:
In this observational prospective studi patients with invasive breast cancer no more than 5 cm and clinically node negative, scheduled for conservative surgery and Sentinel Node Biopsy (SNB), are enrolled in the protocol if they have 1-2 sentinel lymphnodes (SLNs) with macrometastases. SLN status will be checked on definitive sections.

DETAILED DESCRIPTION:
In recent years, breast oncologic surgery has aimed to omit axillary dissection in cases where no more than two sentinel lymph nodes are positive, particularly when complementary radiotherapy to the whole breast is planned.

Radiation therapy to the axillary lymph nodes ensures excellent locoregional control in patients with primary tumor no more than 5 centimeter and 1-2 macrometastatic sentinel lymph nodes, and appears to carry fewer side effects than axillary dissection.

Arm lymphedema is indeed one of the most well-known long-term complications of breast cancer treatment, impacting the quality of life for patients undergoing lymphadenectomy. In this scenario, the study proposes a treatment of hypofractionated intensity-modulated radiotherapy (IMRT) to the breast and axillary lymph nodes with the aim of further containing the risk of developing ipsilateral arm lymphedema. IMRT improves the dosimetric profile of surrounding organs at risk in the treated area, with better dose conformity to the target volume compared to tangential fields used in conventional 3D conformal techniques (as employed in most trials described so far).

ELIGIBILITY:
Inclusion Criteria:

1. Histological proven invasive breast cancer
2. Breast conserving surgery with no axillary dissection
3. Tumor dimension no more then 5 cm and no more than 2 positive sentinel node

5) Negative surgical margin (no tumor cell on ink) 6) Performance Status (PS) <2 7) Age >18 8) Written informed consent

Exclusion Criteria:

1. Previous thoracic RT
2. Mixed connective disorders
3. Distant metastases
4. Severe lung or cardiac diseases
5. Neoadjuvant systemic therapies
6. Axillary dissection
7. No surgical axillary investigation
8. Mastectomy
9. Axillary micrometastasis or isolated tumor cell

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with invasive breast cancer staged clinically node negative and no more then 5 cm of breast tumor, scheduled for quadrantectomy and SNB, are enrolled in the protocol if they have 1-2 SLNs with macrometastases. SLN status will be checked on definitive sections
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-04-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with arm lymphedema | 1 year
  Incidence of ipsilateral arm lymphedema 1 year after the completion of adjuvant radiotherapy

SECONDARY OUTCOMES:
Evaluation of cute locoregional toxicity at breast and axilla | 6 months
  During treatment and within 6 months, acute toxicity is assessed by physician using RTOG scale
Evaluation of chronic toxicity at breast and axilla | 5 years
  Chronic toxicity is evaluated according to LENT-SOMA system as from 6 months onward
Disease free survival | 5 years
  Number of patients with an oncological event (local, regional and distant recurrence free survival)
Overall survival | 5 years
  Number of patient alive after 5 years of follow up
Quality of life (QoL) in order to evaluate pain, itching and burning at breast or axilla | 5 years
  Numeric Rating Scale (NRS) (NRS-11) is an 11-point scale for patient self-reporting of pain. It is used for rating symptoms like pain, itching and burning

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Leonardi, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy